CLINICAL TRIAL: NCT04139382
Title: Using Telemedicine to Improve Early Medical Abortion at Home
Acronym: UTAH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study suspended on 31 March 2020 due to COVID-19 pandemic. Aimed to restart study early 2021, but decision taken to formally terminate the study on 31st August 2021
Sponsor: NHS Lothian (Other Government)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC19076; IRAS (Other: 264265)
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Abortion Early; Abortion in First Trimester
Keywords: Telemedicine; Telephone; Remote

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Telephone Consultation for women requesting abortion
  Interventions: Other: Telephone Consultation
- Control (Active Comparator): Face-to-face consultation for women requesting abortion
  Interventions: Other: Face-to-Face Consultation

INTERVENTIONS:
Other: Telephone Consultation — A telephone consultation comprising clinical history, contraception planning, explanation of medical method of abortion
  Arms: Intervention
Other: Face-to-Face Consultation — A face-to-face consultation comprising clinical history, contraception planning, explanation of medical method of abortion
  Arms: Control

SUMMARY:
The investigators plan a trial comparing telephone consultations for women requesting early medical abortion (EMA - under 10 weeks pregnant) to regular face-to-face consultations.

In Scotland, 7 out of 10 women having an abortion choose EMA. The clinic visit to discuss EMA is lengthy (2-3 hours). Much time is spent between having tests and waiting to consult a doctor or nurse. Women can struggle with time off work or childcare for lengthy daytime appointments.

There is some evidence from other countries that telephone consultations for EMA are a safe and acceptable alternative.

In this study, women seeking EMA will be randomised to face-to-face (standard care) or a planned telephone consultation (in advance of the clinic visit).

The investigators will determine the success of the EMA in both groups, women' satisfaction with the consultation and possible advantages and disadvantages. If telephone consultations prove to be effective and acceptable then this will change EMA provision throughout Scotland.

DETAILED DESCRIPTION:
This study is a randomised controlled trial comparing telephone consultation to face-to-face consultation prior to early medical abortion at home (EMA).

The majority of patients seeking abortion care in NHS Lothian will self-refer by telephone to the Lothian Abortion Referral Service (LARS).

Routinely, patients are asked the date of their last menstrual period (LMP) by administrative staff. They then collect basic contact information and book an appointment to come to clinic within 5-7 days.

For all women who self report an LMP that is less than 10 weeks to the date of the appointment they are offered, the administrative staff at LARS will read a short statement describing the project and ask if the patient is happy to be contacted by a member of the research team to discuss further. If they agree, they will also be directed to the LARS webpage where a copy of the Participant Information Sheet (PIS) will be available. The patient's contact details will be passed to the research nurse or doctor who will then call the patient back.

At call back, the researcher will confirm that the patient has read the PIS and answer any questions and give further information as required. If the patient wishes to participate, verbal consent will be obtained using a standard form.

The patient (now participant) will then be randomised to either the intervention arm (telephone consultation) or standard of care (face-to-face consultation).

For participants in the standard of care arm:

They will attend clinic as usual at the appointment already issued by LARS. After the consultation, they will be asked to complete a questionnaire (either self-administered or researcher-administered) about their preparedness for EMA.

14-20 days later a follow-up questionnaire will be completed with the researcher via telephone, internet or post to assess completion of abortion (using the outcome of a low sensitivity urinary pregnancy test, the standard method used at the abortion service), overall acceptability of consultation and EMA process and what method of contraception they have selected.

For participants in the intervention arm:

They will have a telephone consultation either immediately after they have been randomised or at another point up to the evening before they are due to attend clinic, depending on their preference. The content of the consultation will be identical to that of a face-to-face consultation.

They will attend clinic as planned at their allocated appointment time for an ultrasound scan to confirm gestation, to have standard blood tests and infection screen, complete consent paperwork for their abortion care procedure (as per standard care) and receive their medications.

Before leaving the department, they will be asked to complete a questionnaire (either self-administered or researcher-administered) about their preparedness for EMA.

14-20 days later a follow-up questionnaire will be completed with the researcher via telephone, internet or post to assess completion of abortion (using the outcome of a low sensitivity urinary pregnancy test, the standard method used at the abortion service), overall acceptability of consultation and EMA process and what method of contraception they have selected.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported last menstrual period (LMP) less than 10 weeks on day of appointment
* Self-referral to Lothian Abortion Referral Service (LARS)
* Aged 16 or over at the time of procedure
* Preference for EMA
* Ability to give informed consent

Exclusion Criteria:

* Requires interpreter
* Patient preference for surgical method of abortion

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of medical abortion | 2 weeks after administration of abortion medications (via telephone)
  Complete abortion as assessed by self-performed low-sensitivity urinary pregnancy test

SECONDARY OUTCOMES:
Preparedness for medical abortion | Within 1 week of randomisation (on day of clinic attendance)
  A Likert-scale rating of how prepared participant felt for medical abortion
Satisfaction with consultation | 2 weeks after administration of abortion medications (via telephone)
  A Likert-scale rating of how satisfied participant was with consultation for medical abortion
Contraception | Case note review at 2 weeks
  Rate of uptake of contraceptive methods following consultation
Ineligibility for EMA | Within 1 week of randomisation (on day of clinic attendance)
  Proportion of participants who are not eligible for early medical abortion when they attend clinic for confirmatory ultrasound
Time taken | Within 1 week of randomisation (on day of clinic attendance)
  Time taken in consultation and in clinic
Unscheduled contact | 4 weeks after administration of abortion medications
  Unscheduled contact with abortion service or hospital within 4 weeks of EMA for concern related to EMA

CONTACTS AND LOCATIONS:
Overall Officials: Sharon T Cameron, MD FRCOG, Principal Investigator — University of Edinburgh
Locations (1):
- Chalmers Centre for Sexual and Reproductive Health, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We cannot share individual level data

REFERENCES:
- [Derived] Reynolds-Wright JJ, Norrie J, Cameron ST. Using telemedicine to improve early medical abortion at home (UTAH): a randomised controlled trial to compare telemedicine with in-person consultation for early medical abortion. BMJ Open. 2023 Sep 13;13(9):e073630. doi: 10.1136/bmjopen-2023-073630. PMID 37709327
- [Derived] Reynolds-Wright JJ, Norrie J, Cameron ST. UTAH: Using Telemedicine to improve early medical Abortion at Home: a protocol for a randomised controlled trial comparing face-to-face with telephone consultations for women seeking early medical abortion. BMJ Open. 2021 Jun 16;11(6):e046628. doi: 10.1136/bmjopen-2020-046628. PMID 34135047